CLINICAL TRIAL: NCT00938145
Title: Imaging of Bladder Cancer Using Clinical 3 Tesla MRI and EX-VIVO Ultra-High-Field MRI.
Brief Title: 3 Tesla MRI in Patients With Bladder Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Michael V Knopp MD PhD, Principal Investigator, University of Cincinnati
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OSU-08063; NCI-2012-00937 (Registry Identifier: Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2009-07-10; First posted 2009-07-13 (Estimated); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Bladder Cancer
Keywords: recurrent bladder cancer; stage II bladder cancer; stage III bladder cancer; stage IV bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Drug Therapy; Cystectomy; Lymph Node Excision; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- MRI+surgery (Experimental): 3 Tesla MRI/Cystectomy and Lymphadenectomy/Urinary Diversion/Specimen Ultra-High field MRI
  Interventions: Procedure: Specimen Ultra-High field MRI; Procedure: Cystectomy and Lymphadenectomy
- MRI+surgery+chemotherapy (Experimental): 3 Tesla MRI/Cystectomy and Lymphadenectomy/Urinary Diversion/Specimen Ultra-High field MRI/chemotherapy
  Interventions: Procedure: Specimen Ultra-High field MRI; Drug: chemotherapy; Procedure: Cystectomy and Lymphadenectomy

INTERVENTIONS:
Procedure: Specimen Ultra-High field MRI — Immediately following removal of the bladder and lymph nodes, the specimens will be transported to the ultra-high-field MRI scanner for high resolution imaging.
Drug: chemotherapy — The majority of patients will be candidates to receive neoadjuvant chemotherapy prior to radical cystectomy as part of standard clinical care. Patients will most often receive cisplatin based therapy for a period of three months (four 21 day cycles).
  Other Names: chemo
  Arms: MRI+surgery+chemotherapy
Procedure: Cystectomy and Lymphadenectomy — The patient will undergo radical cystectomy and pelvic lymph node dissection with no deviation from standard surgical care. A urinary tract reconstruction will follow as either a continent or incontinent form of diversion.
  Other Names: surgery

SUMMARY:
RATIONALE: New diagnostic procedures, such as 3 Tesla magnetic resonance imaging (MRI), may help find bladder cancer and learn the extent of disease.

PURPOSE: This clinical trial is studying how well 3 Tesla MRI works in finding cancer in patients with bladder cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate whether 3 Tesla MRI can accurately determine the primary tumor (T) stage and pelvic lymph nodes (N) stage in patients with localized bladder cancer as compared to histopathology staging.

Secondary

* To determine whether 3 Tesla MRI can determine if the primary bladder tumor is responding to neoadjuvant chemotherapy at the mid-point of the planned treatment (after 2 courses).
* To assess whether an ex-vivo ultra-high-field MRI (4.7-11.7 Tesla) tissue scan can more accurately determine clinical stage of a primary bladder tumor and local extent of the disease (i.e., involvement of contiguous organs and regional lymph nodes) as compared to histopathology staging.

OUTLINE: Patients may receive neoadjuvant chemotherapy (typically four 21-day courses of cisplatin-based therapy) followed by standard radical cystectomy and lymph node dissection.

Patients undergo a 3 Tesla MRI scan at baseline to stage the primary tumor, regional lymph nodes, and to rule out distant sites of disease. The MRI includes diagnostic high-resolution anatomical images (e.g., T1-weighted and T2-weighted images along axial or optimal directions) and experimental images including functional MRI (e.g., dynamic contrast-enhanced MRI, diffusion-weighted MRI, MR spectroscopy, and chemical exchange-dependent saturation-transfer imaging). Patients also undergo a 3 Tesla MRI scan after 2 courses of neoadjuvant chemotherapy and after completion of neoadjuvant chemotherapy. Patients not receiving neoadjuvant chemotherapy undergo a 3 Tesla MRI scan 2-4 weeks before radical cystectomy and lymph node dissection.

Specimens from the radical cystectomy and pelvic lymph node dissection are examined ex-vivo by ultra-high-field MRI and the Micro-Imaging Specimen Study Form is completed. The specimens are then examined by the pathology department as per standard routine.

ELIGIBILITY:
Inclusion Criteria:

* Known bladder cancer
* Scheduled for radical cystectomy and lymph node dissection.
* Able and willing to give valid written informed consent.
* No contraindications to the MRI(magnetic resonance imaging).

Exclusion Criteria:

* Not pregnant, planning to become pregnant during the study, or nursing.
* No allergy to contrast agents.
* Patient with significant renal insufficiency, i.e. an estimated glomerular filtration rate(eGRF) less than 30 mL/min/1.73m2.
* Any condition conflict based on the investigation's clinical judgment that would prevent the patient from completion all trial assessments and visits.
* Inability or unwillingness to cooperate with requirements of this trial.
* Patients who exhibit noticeable anxiety and/or claustrophobia or who exhibit severe vertigo when they are moved into the MR.
* Patients with sickle cell anemia and other hemolytic anemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2009-07-08 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Agreement in tumor staging between pathology and 3 Tesla MRI | up to 24 months

SECONDARY OUTCOMES:
Agreement in lymph node staging between pathology and 3 Tesla MRI | up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael V. Knopp, MD, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu